CLINICAL TRIAL: NCT06080750
Title: Potential Role of Inflammasome NLRP3 And IL-1B Gene Expression In COVID-19 Patients: Impact of Ferretin and D -Dimer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Abdel-Baset Ahmed Aly, Pharmacist, Assiut University
Other Study IDs: NLRP3 & IL-1B in covid19
Record Dates: First submitted 2023-10-10; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Inflammasome NLRP3 And IL-1B Gene Expression in COVID-19 Patients
MeSH Terms: interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples With DNA — qRT-PCR: for gene expression of NLRP3 inflammasome and IL-1B in blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy: as a control group
  Interventions: Genetic: Quantitative Real Time Polymerase chain reaction (qRT-PCR); Diagnostic Test: ELISA and colorimeter
- mild to moderate covid-19: mild-moderate symptoms
  Interventions: Genetic: Quantitative Real Time Polymerase chain reaction (qRT-PCR); Diagnostic Test: ELISA and colorimeter
- sever covid-19.: severe symptoms
  Interventions: Genetic: Quantitative Real Time Polymerase chain reaction (qRT-PCR); Diagnostic Test: ELISA and colorimeter

INTERVENTIONS:
Genetic: Quantitative Real Time Polymerase chain reaction (qRT-PCR) — to study gene expression of NLRP3 inflammasome and IL-1B in blood
  Other Names: qRT-PCR
Diagnostic Test: ELISA and colorimeter — IL-6 and total LDH

SUMMARY:
2.1 Study the role of NLRP3 inflammasome in COVID-19 patients. 2.2 Study the gene expression of NLRP3 and IL-1β in blood samples of COVID-19 patients and compare to apparently healthy subjects.

2.3 Correlation between NLRP3, IL-1β, IL-6 and severity of the disease. 2.4 Impact of ferritin and D-dimer on inflammasome componnets NLRP3, IL-1β IL-6 .

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a viral infection that results in respiratory disease, which can evolve into multiorgan failure (MOF), leading to death (Aida A Abdelmaksoud et al., 2021).

The first cases of COVID-19 were detected in Wuhan, China, in 2019. Since then, the illness has spread rapidly around the country and the world reaching a pandemic level (Rocklöv J et al., 2020). Cases have been reported in more than 180 countries to the World Health Organization (WHO), including more than two million deaths (WHO, 2021).

Several biochemical alterations have been described in COVID-19 patients as lymphopenia, thrombocytopenia and increased levels of C-reactive protein. The hallmark of severe COVID-19 is the cytokine storm accompanied by a hyperinflammatory response in the host due to the release of large amounts of pro-inflammatory cytokines IL-1β, IL-6, IL-2, IL-7, TNF-α, interferon-γ (IFN)-γ, CRP, procalcitonin (PCT), lactate dehydrogenase (LDH), erythrocyte sedimentation rate (ESR) and ferritin (Marcello Ciaccio and Agnello, 2020; Shah A., 2020).

The inflammasome is a multiprotein complex, known for its role in the innate immune response against viral diseases and a regulator of processing of the pro-inflammatory cytokines interleukin (IL)-1β and IL-18. Inflammasome contains a NOD-like receptor (NLR) sensor protein and pyrin domain-containing 3 , after which, NLRP3 Inflammasome was named (de Rivero Vaccari et al., 2020). The presence of inflammasome-derived products such as IL-1β, IL-18, and LDH in patients' sera suggests inflammasome engagement (Chen G et al., 2020).

Increased IL-6, IL-10, and IL-4 were found in patients when compared with controls, indicating that SARS-CoV-2 infects human monocytes and triggers NLRP3 inflammasome activation. However, the definitive demonstration of NRLP3 inflammasome participation is still required because these products can be produced via inflammasome-independent pathways (Rodrigues et al., 2021). But, the possible contribution of NLRP3 inflammasome activation and their ability to induce IL-1β production is still not clear .

The pronounced inflammatory characteristics of COVID-19 prompted us to investigate the expression of the NRLP3 inflammasome and its relation to IL-1B in disease development and severity and to determine the best anti-inflammatory will be used in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient aged 18years and over presented to Assiut University Hospital
* Suspected of covid19 because of the presence of symptoms suggestive of pneumonia (fever>38) and at least one of the following symptoms ;cough, dyspnea, tachpnea or hypoxia
* having RT-PCR (confirmed positive PCR)
* Chest CT within 5 days of initial PCR

Exclusion Criteria:

* Cases less than 18 years old
* Cancer patients (affect result of study as they have disrubted level of these biomarker)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Covid 19 patients andcontrol
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
gene expression of NLRP3, IL-1β and level IL-6 | 3 years
  Fold change increased in gene expression of NLRP3, IL-1β and level IL-6 and severity of the disease

SECONDARY OUTCOMES:
ferritin and D-dimer on NLRP3, IL-1β and IL-6 | 3 years
  The relation between level of ferritin and D-dimer on NLRP3, IL-1β and IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Ayat A Sayed, M.D, Study Director — associate professor; Mona A AlBaz, M.D, Study Chair — Professor
Locations (1):
- Biochemistry department,Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdelmaksoud AA, Ghweil AA, Hassan MH, Rashad A, Khodeary A, Aref ZF, Sayed MAA, Elsamman MK, Bazeed SES. Olfactory Disturbances as Presenting Manifestation Among Egyptian Patients with COVID-19: Possible Role of Zinc. Biol Trace Elem Res. 2021 Nov;199(11):4101-4108. doi: 10.1007/s12011-020-02546-5. Epub 2021 Jan 7. PMID 33409924
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] de Rivero Vaccari JC, Dietrich WD, Keane RW, de Rivero Vaccari JP. The Inflammasome in Times of COVID-19. Front Immunol. 2020 Oct 8;11:583373. doi: 10.3389/fimmu.2020.583373. eCollection 2020. PMID 33149733
- [Background] Ciaccio M, Agnello L. Biochemical biomarkers alterations in Coronavirus Disease 2019 (COVID-19). Diagnosis (Berl). 2020 Nov 18;7(4):365-372. doi: 10.1515/dx-2020-0057. PMID 32589600
- [Background] Rocklov J, Sjodin H, Wilder-Smith A. COVID-19 outbreak on the Diamond Princess cruise ship: estimating the epidemic potential and effectiveness of public health countermeasures. J Travel Med. 2020 May 18;27(3):taaa030. doi: 10.1093/jtm/taaa030. PMID 32109273
- [Background] Rodrigues TS, de Sa KSG, Ishimoto AY, Becerra A, Oliveira S, Almeida L, Goncalves AV, Perucello DB, Andrade WA, Castro R, Veras FP, Toller-Kawahisa JE, Nascimento DC, de Lima MHF, Silva CMS, Caetite DB, Martins RB, Castro IA, Pontelli MC, de Barros FC, do Amaral NB, Giannini MC, Bonjorno LP, Lopes MIF, Santana RC, Vilar FC, Auxiliadora-Martins M, Luppino-Assad R, de Almeida SCL, de Oliveira FR, Batah SS, Siyuan L, Benatti MN, Cunha TM, Alves-Filho JC, Cunha FQ, Cunha LD, Frantz FG, Kohlsdorf T, Fabro AT, Arruda E, de Oliveira RDR, Louzada-Junior P, Zamboni DS. Inflammasomes are activated in response to SARS-CoV-2 infection and are associated with COVID-19 severity in patients. J Exp Med. 2021 Mar 1;218(3):e20201707. doi: 10.1084/jem.20201707. PMID 33231615
- [Background] Shah A. Novel Coronavirus-Induced NLRP3 Inflammasome Activation: A Potential Drug Target in the Treatment of COVID-19. Front Immunol. 2020 May 19;11:1021. doi: 10.3389/fimmu.2020.01021. eCollection 2020. No abstract available. PMID 32574259